CLINICAL TRIAL: NCT07141290
Title: Motor Control Enhancement Based on Augmented Feedback Exergame
Brief Title: Motor Control Exergame
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Motor_control_exergame
Record Dates: First submitted 2025-07-21; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-07

CONDITIONS: Proprioception Knee; Healthy Volunteers
Keywords: Home-based exergame; auditory feedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auditory feedback group (Experimental): Participants play the game with auditory feedback
  Interventions: Device: Sound supported fish and bunny game
- Control group (Active Comparator): Participants play the game without auditory feedback
  Interventions: Device: Silent fish and bunny game

INTERVENTIONS:
Device: Silent fish and bunny game — Participants play two levels of a computer game. In one level they need to squat at different levels to make a bunny jump and catch some carrots. In the other level they need to catch fiches by adjusting the extension of their leg.
  Arms: Control group
Device: Sound supported fish and bunny game — In the auditory feedback group sound is used to transfer the Knowledge of Results. The sound is linked to the joint position.
  Arms: Auditory feedback group

SUMMARY:
This study investigates whether auditory feedback improves the performance of people training squats or kicking movement with a computer game that gives feedback on the user's performance.

During the study participants are wearing sensors that record the movement of their upper and lower leg and the muscle activity of the muscles used to perform squatting and kicking. At the beginning of the measurement participants will be asked to perform 10 squats, 10 half squats, and to hold some positions for a short period. Then participants will be allocated to group 1 or group 2 by a draw.

Group 1: plays the exergame without sound Group 2: plays the exergame with sound

Participants play four rounds of a squatting and four rounds of a kicking game. After playing the game they are again asked to perform 10 squats, 10 half squats, and to hold some positions for a short period. Furthermore, they fill a questionnaire in which they indicate whether they liked the game.

The researchers use the measurements taken prior and after the game to see whether participants improved in kicking and squatting. Furthermore they compare which group scores better in the game to see whether auditory feedback helps to understand the game story.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Healthy based on self-report

Exclusion Criteria:

* Pregnancy based on self-report
* Orthopedic problems, musculoskeletal disorder, or prior surgery on the lower extremities based on self-report
* Abuse of drugs, growth hormones, anabolic steroids, or performance enhancing substances based on self-report
* Participants with a known plaster or metal allergy based on self-report
* Not being able to follow the instructions given in Dutch or English
* Not willing to wear shorts/ expose the skin of the legs for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Knee angle error | Baseline and Day1
  The knee angle is defined as the angle between the calibrated coordinate system of the mid-shank and that of the BF of the non-dominant leg measured by means of inertial measurement units. This value is compared to the desired knee angle.

SECONDARY OUTCOMES:
User experience questionnaire (UEQ) | Day 1
  User experience is assessed with the standardized user experience questionnaire (UEQ). The UEQ is a stnadardized 26 item questionnaire which assesses the dimensions Attractiveness, Perspicuity, Efficiency, Dependability, Stimulation and Novelty. For each question the participant answers on a 7 point Likert scale. The maximum number of points is 128. The minimum number of points is 26.
Muscle activity and coordination | baseline and Day1
  Electromyography data was accumulated from the major muscles in the leg. These were analyzed using NMF to see whether activation patterns are different depending on the presence of auditory feedback.
Motivation | Day1
  Motivation of the participants during game play is assessed with the standardized Intrinsic Motivation Inventory (IMI) questionnaire. The version that is used within this study has 22 questions. The questions are answered on 7 point likert scales. The minimum score is 22. The maximum score is 154.
In game performance | baseline and Day 1
  In game performance is measured by comparing scores participants get in the game.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No